CLINICAL TRIAL: NCT06690619
Title: Effects of Alpha-GPC on Muscle Power, GH Levels, and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: NNB Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NNB-001-012024
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Cognition - Other; Strength Outcomes
Keywords: Cognition; Mental Acuity; Performance; Nootropic; Mental; Acute supplementation

STUDY DESIGN:
Intervention Model Description: N/A. Full detail provided in Study Description
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistical analysis was masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Low Dose Alpha-GPC (Active Comparator): 315 mg dose of alpha-glycerylphosphorycholine (alpha-GPC)
  Interventions: Dietary Supplement: 315 mg Alpha-GPC
- High Dose Alpha-GPC (Active Comparator): 630 mg dose of alpha-glycerylphosphorycholine (alpha-GPC)
  Interventions: Dietary Supplement: 630 mg Alpha-GPC

INTERVENTIONS:
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo
Dietary Supplement: 315 mg Alpha-GPC — 350 mg of 90% pure alpha-GPC (315 mg)
  Arms: Low Dose Alpha-GPC
Dietary Supplement: 630 mg Alpha-GPC — 700 mg of 90% pure alpha-GPC (630 mg)
  Arms: High Dose Alpha-GPC

SUMMARY:
Purpose: To determine the effects of low dose and high dose Alpha-GPC on cognitive performance, muscle performance, and serum growth hormone levels.

Design: Randomized, three-arm, within-subject crossover

Study Participants: 21 apparently healthy men to be recruited at a single investigational center in Northeast Ohio

4 Study Visits

Study Visit 1: Participants will be screened for participation (i.e., medical history, routine blood work, background baseline diet)

Study Visit 2: Participants will ingest one of three supplements (a low dose α-GPC, a high dose α-GPC, or a placebo). Subjects will complete visual analog scale (VAS) questionnaires (assessing mood, motivation, alertness, and concentration) and a cognitive battery (Stroop, Flanker, and N-Back tests) 60 min post ingestion and approximately 3 hours post-ingestion, undergo upper body and lower body power testing and a lower body bout of moderate-intensity exercise 90 min post-ingestion. Also, subjects will undergo blood draws for levels of growth hormone at baseline (prior to supplementation) and 5, 15, 30, and 60 min post lower body bout of exercise. Vital signs and comprehensive side effect profile/ adverse event monitoring will take place throughout the duration of the study. The study will be conducted following ICH-GCP guidelines to ensure subject safety and scientific integrity of the data.

Study Visit 3 and 4 Identical to visit 2 with exception of different supplementation being provided. Supplement administration was randomized using a Latin square approach to reduce variability and enhance statistical power

Primary Outcomes: Upper and lower body peak force production, peak power production, and peak velocity

Secondary Outcomes: Cognitive performance on the Stroop test, Flanker, and N-Back test, serum growth hormone levels, mood, motivation, alertness, and concentration (as assessed by visual analog scales).

Tertiary/Safety Outcomes: Vital signs, side effect profile/AE monitoring

DETAILED DESCRIPTION:
DIET:

* All subjects will be asked to maintain their usual dietary habits throughout the study.
* At screening, all subjects will complete a 24-hour diet recall from the day prior while refraining from any nutrients that might affect choline.
* To replicate screening conditions as closely as possible, subjects will follow their previously recorded 24-hour diet record and fast for 8 hours prior to each laboratory visit.
* An online application (Nutritionix) will be used to analyze their dietary consumption.

BLOODWORK:

•Blood draws will take place during each laboratory visit, and they will be performed by a study nurse or phlebotomist. At screening a single blood draw will be performed with a total blood volume of approximately 12 mL. During visits 2-4 serial blood draws will be performed before and 5-, 15-, 30-, and 60-min post ingestion of the investigational product. During visits 2-4, an intra-venous catheter (flexible tubing to enable blood sampling) will be inserted into an upper extremity vein. Blood samples will be collected up to 5 times over 4 hours.

EXERCISE TRAINING AND PHYSICAL ACTIVITY CONTROL

•Subjects will be asked to maintain their activities of daily living and abstain from exercise for 48 hours prior to each trial.

TEST PRODUCTS

* After qualifying for the study, subjects will be randomly assigned to receive a placebo, a low dose of α-GPC, and a high dose of α-GPC using a Latin Square design.

  * Low dose of α-GPC (350 mg)
  * High dose of α-GPC (700 mg)
  * Placebo (containing maltodextrin)
* Supplements will be provided in identical-looking capsules with label directions and Study Protocol Number.
* Subjects will consume each supplement in the presence of the medical staff.
* There will be no less than one week between each trial, though this may be longer depending on scheduling.
* As stated earlier, subjects who withdraw from the study prior to completing all three trials may be replaced.

DETAILED STUDY PROCEDURES

Visit 1 (Screening)

* Medical history, safety blood work (CBC, CMP, and Lipid Panel)
* Body composition (bioimpedance-BIA)
* Baseline diet (24hr recall).
* Body weight
* Familiarization trial for the cognitive battery (Stroop, Flanker, and N-Back test).

Visits 2-4

* Subjective feelings of mood, motivation, alertness, and concentration will be assessed 60 minutes post ingestion and approximately 3 hours post-ingestion. All assessments will be made using 100 mm anchored visual analogue scales (VAS).
* Three repetitions of the Stroop (2-min tests), Flanker, and N-Back (90s tests) tests will be assessed 60 minutes post ingestion and approximately 3 hours post-ingestion.

  * Stroop - https://www.psytoolkit.org/lessons/stroop.html
  * Flanker - https://www.psytoolkit.org/experiment-library/flanker.html
  * N-Back - https://www.lumosity.com/app/v4/games/speed-match-overdrive-web
* Upper and lower body muscular power will be assessed with a Tendo unit. For the upper body, the bench press throw using a submaximal load (i.e., 50% of 1RM) will be performed on a Smith machine. For the lower body, a vertical jump will be performed. Both tests will be performed 90 minutes post-ingestion.
* Moderate intensity lower body exercise bout consisting of 6 sets of 10 repetitions at 70% of 1RM of squats using a metronome for cadence (15 reps per min) on a Smith machine approximately 2 hours post-ingestion.
* Growth hormone will be measured via blood draw before supplementation ingestion and 5, 15, 30, and 60 min post lower body exercise bout.
* Body weight
* Vital signs will be assessed prior to supplementation, 60 minutes post ingestion, and approximately 3.5 hr post-ingestion.

Study Schematic:

Informed Consent: Visit 1 Inclusion/Exclusion Criteria: Visit 1 Medical History: Visit 1 Height, weight, and BMI: Visits 1, 2, 3, 4 24-hr Dietary recall: Visit 1 CBC, CMP, Lipid Panel: Visit 1 Vitals (HR and BP): Visit 1 Bioimpedance Analysis (BIA) for percent body fat: Visit 1 Bench Press Throw for Upper Body Power (Tendo) @ 50%1RM approximately 90 minutes post-ingestion: Visits 2, 3, 4 Vertical Jump for Lower Body Power (Tendo) approximately 90 minutes post-ingestion: Visits 2, 3, 4 Lower body exercise bout consisting of squats on a Smith machine (6 x 10 @70%1RM) beginning approximately 2 hours post-ingestion: Visits 2, 3, 4 Cognitive performance battery (N-back, Flanker, Stroop) (60 min post ingestion and approximately 3 hours post-ingestion on visits 2-4 only): Visits 1, 2, 3, 4 Serum GH (before ingestion and 5, 15, 30, and 60 min post lower body exercise bout): Visits 1, 2, 3, 4 VAS (mood, motivation, alertness, and concentration) 60 min post ingestion and approximately 3 hours post-ingestion): Visits 2, 3, 4 Vitals (HR and BP) monitoring (at baseline, 60 min post ingestion, and approximately 3.5 hours post-ingestion): Visits 2, 3, 4 24 hr Diet Records/Analysis/Repeat: Visits 2, 3, 4 Protocol Compliance (diet and physical activity log check): Visits 2, 3, 4 Dispense Test Product: Visits 2, 3, 4 Adverse Events Monitoring: Visits 1, 2, 3, 4

METHODS AND INSTRUMENTATION:

* Health history will be determined using a standardized (IRB-approved) questionnaire.
* Heart rate and blood pressure will be measured using an automated sphygmomanometer.
* Body composition will be measured using a bioimpedance device (InBody 570- https://inbodyusa.com/products/inbody570/).
* Standing height will be determined using a wall-mounted stadiometer.
* Body weight and height will be measured using a Seca Medical Scale (https://www.hogentogler.com/seca/769-physician-scale.asp?gclid=EAIaIQobChMIxoqxi6ef8wIVtmpvBB34QAwzEAQYAyABEgIVIPD_BwE).
* Upper and lower body muscular power will be determined using a Tendo power analyzer (Tendo Sport- https://www.tendosport.com/products/tendo-unit/overview/)
* A Central Lab (LabCorp, Dublin, OH) will be utilized to transport and analyze all blood samples.
* Diet records will be analyzed using the online application (Nutritionix).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between 25 and 55 years (inclusive).
* Body Mass Index of 18.5-34.9 (inclusive).
* Body weight of at least 120 pounds.
* Resistance training history of at least 2 years.
* Normotensive (supine, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg.
* Normal supine, resting heart rate (< 90 per minute).
* Willing to duplicate their previous 24-hour diet, refrain from alcohol and caffeine for 24 hr prior to each trial, refrain from exercise 48 hr prior to each trial, refrain from any nutrients that might affect choline 24 hr prior to each trial, and fast for 8 hours prior to each trial.

Exclusion Criteria:

* Highly trained or competitive athletes.
* History of diabetes, asthma, gout, fibromyalgia or clinical diagnosis of IBS/IBD.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* History of psychiatric disorder.
* History of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Use of any dietary supplements that may confound the study or its endpoints, including creatine, BCAA, HMB, betaine, beta-alanine, etc.
* Use of stimulants or anxiety or ADHD medication.
* Caffeine intake of three or more cups of coffee or equivalent (>400 mg) per day.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence.
* Smokers.
* Clinically significant abnormal laboratory results at screening.
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition or disease (e.g., rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Concomitant use of corticosteroids or testosterone replacement therapy (ingestion, injection, or transdermal).
* Known allergy or sensitivity to any ingredient in the test formulations as listed in the Certificates-of-Analysis.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoint or place the subject at increased risk of harm if they were to participate.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance-NBack | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during visits 2, 3, and 4
  The N Back cognitive performance test (https://www.lumosity.com/app/v4/games/speed-match-overdrive-web )
Cognitive Performance | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during visits 2, 3, and 4
  Flanker Cognitive Performance Test (https://www.psytoolkit.org/experiment-library/flanker.html)
Cognitive Performance | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during visits 2, 3, and 4
  Stroop Color Matching Test

SECONDARY OUTCOMES:
Lower Body Power | Assessed 90 minutes post-ingestion during each study visit
  Vertical Jump for Lower Body Power (Tendo)
Upper Body Power | Assessed 90 minutes post-ingestion during each study visit
  Bench Press Throw for Upper Body Power (Tendo) @ 50%1RM
Growth Hormone | Assessed before exercise and 5, 15, 30, and 60 minutes after exercise during visits 2, 3, and 4
  Serum Growth Hormone Concentrations
Perceived mood assessed using visual analog scale | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during visits 2, 3, and 4
  Perceived mood assessed using the Visual Analog Scale (VAS), a 0-100 scale where 0 indicates 'worst mood imaginable' and 100 indicates 'best mood imaginable.' Higher scores represent better perceived mood.
Perceived motivation assessment using visual analog scales | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during visits 2, 3, and 4
  Perceived motivation assessed using the Visual Analog Scale (VAS), with a range of 0-100 where 0 indicates 'no motivation' and 100 indicates 'maximum motivation.' Higher scores represent better perceived motivation.
Perceived Alertness Assessment Using Visual Analog Scale (VAS) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during visits 2, 3, and 4
  Perceived alertness assessed using the Visual Analog Scale (VAS), with a range of 0-100 where 0 indicates 'no alertness' and 100 indicates 'maximum alertness.' Higher scores represent better perceived alertness.
Perceived Concentration Assessment Using Visual Analog Scale (VAS) | Assessed 60 minutes after ingestion of assigned test product and approximately 3 hours after ingestion during visits 2, 3, and 4
  Perceived concentration assessed using the Visual Analog Scale (VAS), with a range of 0-100 where 0 indicates 'no concentration' and 100 indicates 'maximum concentration.' Higher scores represent better perceived concentration.
Non-exertional Heart Rate Measurement | Assessed 60 minutes after ingestion of assigned test product and approximately 3.5 hours after ingestion during visits 2, 3, and 4
  Heart rate measured in a non-exertional state using an automated sphygmomanometer.
Non-exertional Blood Pressure Measurement (Systolic and Diastolic) | Assessed 60 minutes after ingestion of assigned test product and approximately 3.5 hours after ingestion during visits 2, 3, and 4
  Blood pressure measured in a non-exertional state using an automated sphygmomanometer. Both systolic and diastolic pressures will be assessed.

OTHER OUTCOMES:
Percent Body Fat | At baseline (Visit 1), at the start of the study.
  Percent body fat assessed using bioelectrical impedance analysis
Dietary Intake | Day 1, Day 8, and Day 15
  24-Hour Dietary Intake using 24-hour recall approach. Energy and macronutrient intake were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Ziegenfuss, PhD, Principal Investigator — Center for Applied Health Sciences
Locations (1):
- Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- [Derived] Kerksick CM. Acute Alpha-Glycerylphosphorylcholine Supplementation Enhances Cognitive Performance in Healthy Men. Nutrients. 2024 Dec 9;16(23):4240. doi: 10.3390/nu16234240. PMID 39683633